CLINICAL TRIAL: NCT02833584
Title: Safety of Paracetamol as Antipyretic in Treatment of Dengue Infection in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMED2016
Record Dates: First submitted 2016-06-21; First posted 2016-07-14 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Dengue; Transaminitis
Keywords: Paracetamol
MeSH Terms: conditions — Dengue | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Experimental): Eligible patients will be randomised to receive Paracetamol prn for fever at maximum dosage of 500 mg PO q 4 hr (3 gm/day)
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): Eligible patients will be randomised to receive Placebo prn for fever at maximum dosage of 500 mg PO q 4 hr (3 gm/day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — Paracetamol 500 mg x 1 tablets according to patient's body weight
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Placebo — Placebo 500 mg x 1 tablets according to patient's body weight
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether regular dosage of paracetamol causes transaminitis (hepatitis) and evaluate its potency in the treatment of dengue infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 years
* Dengue infection diagnosed by NS1 antigen, Dengue immunoglobulin M antibody, or polymerase chain reaction
* Admitted to the hospital
* Written informed consent from patient or attending relative able to and willing to give informed consent

Exclusion Criteria:

* Other possible cause of fever other than dengue infection
* Pregnancy
* Unable to take medication
* Aminotransferase level above 3 times upper normal limit
* Allergy to paracetamol or tramadol
* Paracetamol indicated for condition other than dengue infection
* Critically ill patient who need ICU or invasive ventilation support
* History of cirrhosis
* Unable to comunicate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with abnormal serum transaminase levels on the last day of fever | Day 1-8
  Serum alanine transaminase and aspartate transaminase level will be measured at admission, and on every morning afterwards until the subject is discharged. The proportion of subjects with abnormal serum transaminase levels will be compared.
Mean serum transaminase level | Day 1-8
  Mean serum transaminase level will be compared.
Mean change in serum transaminase levels | Day 1-8
  The change in serum transaminase levels from baseline at admission will be compared.

SECONDARY OUTCOMES:
Body temperature | 8 days
  Axillary temperature will be recorded every 4 hours until discharge or 8 days after admission, whichever comes first.
Duration of fever | 8 days
  Duration from the fever onset to the last febrile temperature will be compared.
Length of stay | 10 days
  Duration from hospital admission to discharge will be compared.
Number of drug tablet used | 8 days
  Number of drug tablet used will be compared, both paracetamol/placebo and tramadol.

CONTACTS AND LOCATIONS:
Overall Officials: Dhitiwat Changpradub, MD, Study Director — Phramongkutklao College of Medicine and Hospital
Locations (3):
- Thailand (3):
  - Phramongkutklao College of Medicine and Hospital, Bangkok
  - Fort Adisorn Hospital, Changwat Sara Buri
  - Anandamahidol Hospital, Lopburi

REFERENCES:
- [Derived] Vasikasin V, Rojdumrongrattana T, Chuerboonchai W, Siriwiwattana T, Thongtaeparak W, Niyasom S, Lertliewtrakool N, Jitsiri S, Changpradub D. Effect of standard dose paracetamol versus placebo as antipyretic therapy on liver injury in adult dengue infection: a multicentre randomised controlled trial. Lancet Glob Health. 2019 May;7(5):e664-e670. doi: 10.1016/S2214-109X(19)30032-4. PMID 31000133